CLINICAL TRIAL: NCT06239051
Title: Humanitas Fertility Center: The Green (R)Evolution
Brief Title: Greening the Humanitas Fertility Center: How to Build a More Sustainable Medical Daily Routine
Acronym: Green
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: Green Project
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Sustainability; Female Infertility
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to redefine an everyday clinical routine at the Humanitas Fertility center calculating the effects derived from the reduction of inappropriate and avoidable tests, procedures, tools and treatments currently used.

Anonymized patients data about clinical procedures are used, taken from the internal database of the Humanitas fertility center

ELIGIBILITY:
All outpatient, surgical and laboratory procedures, considered as daily clinical routine at the Humanitas Fertility center, will be taken into account, analysed and defined as appropriate or not.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All outpatient, surgical and laboratory procedures, considered as daily clinical routine at the Humanitas Fertility center, will be taken into account, analysed and defined as appropriate or not.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-24 (Actual)

PRIMARY OUTCOMES:
Reduction of avoidable procedures and assessment of its enviromental impact | From 18th September 2023 to 24th September 2023
  Redefine an everyday clinical routine at the Humanitas Fertility center, calculating the effects derived from the reduction of inappropriate and avoidable tests, procedures, tools and treatments currently used

CONTACTS AND LOCATIONS:
Overall Officials: Michele Tedeschi, Study Chair — Humanitas Research Hospital IRCCS, Rozzano-Milan; Paolo Emanuele Levi Setti, Study Director — Humanitas Research Hospital IRCCS, Rozzano-Milan; Camilla Ronchetti, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy